CLINICAL TRIAL: NCT00678067
Title: Effects of Docosahexaenoic Acid (DHA) and Eicosapentaenoic Acid(EPA)Supplementation on DHA Plasmatic Status and Blood Lipid Profile in Hypercholesterolemic Children in Addition to National Cholesterol Education Program Step I Diet
Brief Title: Effects of Docosahexaenoic and Eicosapentaenoic Acids in Hypercholesterolemic Children Plus Diet on Docosahexaenoic Acid (DHA) Status
Acronym: DHA-RICHOIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Silvia Decarlis, MD, Dept. of Pediatrics, San Paolo Hospital, University of Milan, Italy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DHA-RICH1
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemic children; Docosahexaenoic acid; Eicosapentaenoic acid; Blood lipid profile
MeSH Terms: conditions — Hypercholesterolemia | interventions — Docosahexaenoic Acids; wheat germ oil; Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): 12 hypercholesterolemic children 3-13 years of age
  Interventions: Dietary Supplement: Germ oil; Other: National Cholesterol Education Program (NCEP) Step I Diet
- DHA+EPA group (Experimental): 12 hypercholesterolemic children 3-13 years of age
  Interventions: Dietary Supplement: Docosahexaenoic acid (DHA)+ Eicosapentaenoic acid (EPA); Other: National Cholesterol Education Program (NCEP) Step I Diet
- DHA Group (Experimental): 12 hypercholesterolemic children 3-13 years of age
  Interventions: Dietary Supplement: Docosahexaenoic acid; Other: National Cholesterol Education Program (NCEP) Step I Diet

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid — Soft capsules 500 mg/each; 1 capsule/day for 4 months
  Other Names: DHA
  Arms: DHA Group
Dietary Supplement: Docosahexaenoic acid (DHA)+ Eicosapentaenoic acid (EPA) — Soft capsules, 228 mg DHA + 208 mg EPA /each; 1 capsule/day for 4 months
  Other Names: DHA and EPA mixture
  Arms: DHA+EPA group
Dietary Supplement: Germ oil — Soft capsules, 275 mg linoleic acid + 35 mg linolenic acid + 65 mg oleic acid /each; 1 capsule/day for 4 months
  Other Names: wheat germ oil
  Arms: Placebo
Other: National Cholesterol Education Program (NCEP) Step I Diet — Dietary counselling aimed at achieving NCEP Dietary Guidelines: Total fat intake <30% of total calories, Saturated fat intake <10% of total calories, Polyunsaturated fat intake up to 10% of total calories, monounsaturated fat intake 10-15% of total calories
  Other Names: Dietary intervention; Dietary recommendations

SUMMARY:
To examine whether Docosahexaenoic Acid (DHA) and Docosahexaenoic + Eicosapentaenoic Acids (DHA+EPA) supplementation in addition to National Cholesterol Education Program Step I Diet in Hypercholesterolemic Children increases Docosahexaenoic Acid (DHA) plasma levels in the 2 intervention groups versus placebo. Secondary outcome measure: effect of DHA and DHA+EPA supplementation on blood lipid profile

DETAILED DESCRIPTION:
In a double-blind placebo-controlled trial 36 hypercholesterolemic children, 3-13 years of age, 19 males and 17 females were put on National Cholesterol Education Program (NCEP)Step-I diet and randomised into 3 groups to receive 500 mg/day of purified Docosahexaenoic Acid (DHA), Docosahexaenoic Acid plus Eicosapentaenoic Acid (DHA+EPA) mixture (228 + 208 mg/day respectively), or wheat germ oil as placebo. They underwent at baseline and after a 4 month treatment: EPA and DHA levels in total plasma and in phospholipids, triglycerides, cholesteryl esters; dietary habits by food frequency questionnaire; blood lipid profile (total cholesterol, HDL cholesterol, triglycerides levels)

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary hypercholesterolemia (total cholesterol levels > 200 mg/dl before entering the study)
* BMI >3°and < 97° percentile for age
* First referring to our Lipid Clinic

Exclusion Criteria:

* Secondary dyslipidemia
* Obesity
* Step I diet or any dietary supplement before entering the study

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2005-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Plasma Docosahexaenoic Acid (DHA) levels in DHA group and DHA+EPA group versus placebo after intervention | 4 months

SECONDARY OUTCOMES:
Blood lipid profile variation in DHA Group and DHA+EPA Group versus placebo group after intervention | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Decarlis, MD, Principal Investigator — Dept. of Pediatrics, San paolo Hospital, University of Milan, Italy

REFERENCES:
- [Derived] Verduci E, Agostoni C, Radaelli G, Banderali G, Riva E, Giovannini M. Blood lipids profile in hyperlipidemic children undergoing different dietary long chain polyunsaturated supplementations: a preliminary clinical trial. Int J Food Sci Nutr. 2014 May;65(3):375-9. doi: 10.3109/09637486.2013.858239. Epub 2013 Nov 14. PMID 24228803